CLINICAL TRIAL: NCT04523207
Title: A Multi-center, Open-label, Single-arm Phase 2 Study of the Adjuvant Treatment of Apalutamide and Androgen Deprivation Therapy (ADT) in Treatment-naïve Participants Who Have Undergone Radical Prostatectomy (RP) for Non-metastatic Prostate Cancer and Who Are at High Risk for Metastases
Brief Title: A Study of Apalutamide (Adjuvant Treatment) and Androgen Deprivation Therapy (ADT) in Participants Who Have Undergone Radical Prostatectomy (RP) for Non-metastatic Prostate Cancer and Who Are at High Risk for Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108875; 56021927PCR2041 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apalutamide + Androgen Deprivation Therapy (ADT) (Experimental): In the main study, participants will receive apalutamide 240 milligram (mg) once daily orally along with ADT for 12 cycles (Each cycle is of 28 days). Participants who enrolled in the sub-study will receive apalutamide 240 mg once daily along with relugolix (a type of ADT) 120 mg once daily following a loading dose of 360 mg relugolix orally. Sub-study participants will be receiving relugolix up to Day 28 after which they will be transitioned into the main study from Cycle 2 Day 1 and will continue to receive conventional or oral ADT.
  Interventions: Drug: Apalutamide; Drug: ADT; Drug: Relugolix

INTERVENTIONS:
Drug: Apalutamide — Participants will receive apalutamide 240 mg (4 tablets of 60 mg each) oral tablets during the main study and sub-study.
  Other Names: JNJ-56021927
Drug: ADT — Participants will receive ADT intramuscular or subcutaneously during the main study.
Drug: Relugolix — Participants will receive 120 mg of relugolix following a loading dose of 360 mg of (3 tablets of 120 mg each) relugolix during the sub-study.

SUMMARY:
Main Study: The purpose of main study is to assess if the combination of apalutamide and androgen deprivation therapy (ADT) in participants with high-risk localized prostate cancer improves the biochemical recurrence (BCR) free rate.

Sub-study: The purpose of the sub-study is to assess if the co administration of apalutamide and relugolix is able to maintain castrate levels of testosterone.

ELIGIBILITY:
Inclusion Criteria:

* A candidate for radical prostatectomy (RP) or status post RP. Eligible to receive study intervention between Day 29 and Day 90 post-RP. Post RP prostate-specific antigen (PSA) of <= 0.2 nanograms per milliliter (ng/mL). Has not received other treatment for prostate cancer
* Have recovered from RP procedure and have had no worsening in cardiac risk in the peri-operative period per the clinical judgement of the investigator
* Adequate organ function (hepatic, renal, hematologic and cerebral) determined at the discretion of the treating physician
* Eastern Cooperative oncology Group (ECOG) Performance Status Score of 0 or 1
* Histologically confirmed adenocarcinoma of the prostate and categorized as high risk for recurrent prostate cancer. High risk can be defined based on PSA alone or biopsy or RP specimen as follows: PSA greater than or equal to (>=) 20 ng/ml or; Gleason Score >= 9 in any core on biopsy or; Gleason Score >= 8 (4+4 or 5+3) in greater than (>) 80 percentage (%) of 2 cores on biopsy or; Gleason Score = 8 (4+4 or 5+3) in 1 core as long 5 or more other cores with minimum Gleason Score of 4+3 on biopsy. The determination of high risk may be based on pathology report of biopsy or equivalent criteria from radical prostatectomy

Exclusion Criteria:

* History or presence of soft tissue/bone metastasis or metastasis in distant lymph nodes (pelvic lymph nodes below the iliac bifurcation that are less than (<) 2 centimeter (cm) in diameter [short axis] either radiographically or pathologically are allowed.)
* History of bilateral orchiectomy
* Received an investigational intervention <= 4 weeks before the planned first dose of study intervention
* History of seizure or any condition that in the opinion of the investigator may predispose to seizure or treatment with drugs known to lower the seizure threshold within 4 weeks prior to starting treatment with apalutamide
* Allergy or hypersensitivity to apalutamide, or excipients, unable or unwilling to take androgen deprivation therapy (ADT)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (31):
- United States (31):
  - Arizona Urology Specialists, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Skyline Urology, Sherman Oaks, California
  - Genesis Research, Torrance, California
  - The Urology Center of Colorado, Denver, Colorado
  - Foothills Urology - Golden Off, Lakewood, Colorado
  - Urological Research Network, Hialeah, Florida
  - Idaho Urologic Institute, Meridian, Idaho
  - First Urology, PSC, Jeffersonville, Indiana
  - The Iowa Clinic, West Des Moines, Iowa
  - Wichita Urology Group, Wichita, Kansas
  - Ochsner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Michigan Institute of Urology, PC, Troy, Michigan
  - Adult Pediatric Urology & Urogynecology, P.C, Omaha, Nebraska
  - New Jersey Urology LLC, Voorhees Township, New Jersey
  - Great Lakes Physician PC d/b/a Western New York Urology Associates, Cheektowaga, New York
  - Associated Medical Professionals, Syracuse, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Lancaster Urology, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Lexington Urology, West Columbia, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology Of Virginia, Pllc, Virginia Beach, Virginia
  - Spokane Urology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Shore N, Hafron J, Saltzstein D, Brown G, Belkoff L, Aggarwal P, Phillips J, Bhaumik A, McGowan T. Apalutamide for High-Risk Localized Prostate Cancer Following Radical Prostatectomy (Apa-RP). J Urol. 2024 Nov;212(5):682-691. doi: 10.1097/JU.0000000000004163. Epub 2024 Aug 1. PMID 39088398
- [Derived] Brown G, Belkoff L, Hafron JM, Saltzstein DR, Potdar R, Bhaumik A, Phillips J, McGowan T, Shore ND. Coadministration of Apalutamide and Relugolix in Patients with Localized Prostate Cancer at High Risk for Metastases. Target Oncol. 2023 Jan;18(1):95-103. doi: 10.1007/s11523-022-00932-8. Epub 2022 Dec 6. PMID 36472728

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of main study (12 treatment cycles) and sub study (single treatment cycle). Each cycle was of 28 days. Unique participants were enrolled either into main or sub-study. Study treatment was initiated between Day 29 and 90 post radical prostatectomy. After sub-study completion and serum testosterone assessment (primary analysis) and safety (secondary analysis), participants were transitioned into main study from Cycle 2 Day 1 and continued treatment through Cycle 12 in main study.
Groups:
- Main Study: Apalutamide Plus Androgen Deprivation Therapy (ADT): In main study, participants received apalutamide 240 milligrams (mg; 4 tablets of 60 mg) orally once daily (QD) along with ADT intramuscular or subcutaneous injection from Cycle 1 Day 1 up to Cycle 12. Each cycle was of 28 days.
- Sub Study: Relugolix Followed by Apalutamide Plus Relugolix: In sub-study, participants received a loading dose of relugolix 360 mg (3 tablets of 120 mg) on Day -14 and then relugolix 120 mg orally QD up to Day 28 and accompanied by apalutamide 240 mg (4 tablets of 60 mg tablets) orally QD from Day 1 up to Day 28. Upon completion of 28-day sub-study, participants were transitioned into the main study from Cycle 2 Day 1 and continued to receive apalutamide with ADT (oral relugolix) through Cycle 12. Each cycle was of 28 days.
Period: Overall Study
Arm/Group | Main Study: Apalutamide Plus Androgen Deprivation Therapy (ADT) | Sub Study: Relugolix Followed by Apalutamide Plus Relugolix
Started | 96 | 12
Sub-study Participants Who Completed and Transitioned to Main Study | 0 (Not applicable for the main study.) | 12
Completed | 78 | 9 (Transitioned sub-study participants who completed the main study.)
Not Completed | 18 | 3
Not completed — Adverse Event | 5 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Progressive Disease | 2 | 1
Not completed — Other | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Apalutamide Plus Androgen Deprivation Therapy (ADT) | Sub Study: Relugolix Followed by Apalutamide Plus Relugolix | Total
Number analyzed (Participants) | 96 | 12 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (7.33) | 64.6 (8.46) | 65.2 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 96 | 12 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 87 | 12 | 99
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 2 | 15
  White | 80 | 8 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 96 | 12 | 108

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Biochemical Recurrence (BCR)-Free Rate at Month 24
Description: Confirmed BCR-free rate was estimated from primary efficacy variable, time to confirmed BCR. This was measured as the interval between the date of the first dose of study drug and the date of the first occurrence of confirmed prostate specific antigen (PSA) greater than (>) 0.2 nanogram per milliliter (ng/mL). Confirmation of the PSA value was conducted within 3 to 4 weeks, regardless of study visit and timing. Participants without confirmed PSA > 0.2 ng/mL (including those who were lost to follow-up) were censored on their last PSA measurement date during the treatment phase of the study.
Time Frame: At Month 24
Population: Modified intent-to-treat (MITT) analysis set included all participants who were enrolled in the study, received at least 1 dose of apalutamide, and had a baseline prostate-specific antigen (PSA) and at least 1 post-treatment PSA assessment. Data for this outcome measures was planned to be collected and analyzed for combined population of main study and sub-study (after the participants transitioned into main study).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Apalutamide Plus ADT (Main Study) + Relugolix Followed by Apalutamide Plus Relugolix (Sub Study): In main study, participants received apalutamide 240 milligrams (mg; 4 tablets of 60 mg) orally once daily (QD) along with ADT from Cycle 1 Day 1 up to Cycle 12. In sub-study, participants received a loading dose of relugolix 360 mg (3 tablets of 120 mg) on Day -14 and then relugolix 120 mg orally QD up to Day 28 and followed by apalutamide 240 mg (4 tablets of 60 mg tablets) orally QD from Day 1 up to Day 28. Upon completion of 28-day sub-study, participants were transitioned into the main study from Cycle 2 Day 1 and continued to receive apalutamide along with ADT (of investigator's choice) through Cycle 12. Each cycle was of 28 days.
Arm/Group | Apalutamide Plus ADT (Main Study) + Relugolix Followed by Apalutamide Plus Relugolix (Sub Study)
Number analyzed (Participants) | 108
Percentage of participants | 100 [93.4 to 100]

2. Primary Outcome: Sub-study: Percentage of Participants Who Maintained Testosterone Level Less Than (<) 50 Nanograms Per Deciliter (ng/dL) Through Day 28
Description: Percentage of participants maintaining testosterone level <50 ng/dL through Day 28 were reported.
Time Frame: From Day -14 through Day 28
Population: MITT analysis set included all participants were enrolled in the study, received at least 1 dose of apalutamide, and had a baseline PSA and at least 1 post-treatment PSA assessment. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for main study.
Measure: Number; unit: Percentage of participants
Arm/Group | Sub Study: Relugolix Followed by Apalutamide Plus Relugolix
Number analyzed (Participants) | 11
Percentage of participants | 100

3. Secondary Outcome: Confirmed Biochemical Recurrence (BCR)-Free Rate at Month 12
Description: Confirmed BCR-free rate was estimated from primary efficacy variable, time to confirmed BCR. This was measured as the interval between the date of the first dose of study drug and the date of the first occurrence of confirmed PSA >0.2 ng/mL. Confirmation of the PSA value was conducted within 3 to 4 weeks, regardless of study visit and timing. Participants without confirmed PSA > 0.2 ng/mL (including those who were lost to follow-up) were censored on their last PSA measurement date during the treatment phase of the study.
Time Frame: At Month 12
Population: MITT analysis set included all participants were enrolled in the study, received at least 1 dose of apalutamide, and had a baseline PSA and at least 1 post-treatment PSA assessment. Data for this outcome measures was planned to be collected and analyzed for combined population of main study and sub-study (after the participants transitioned into main study).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Apalutamide Plus ADT (Main Study) + Relugolix Followed by Apalutamide Plus Relugolix (Sub Study)
Number analyzed (Participants) | 108
Percentage of participants | 100 [94.8 to 100]

4. Secondary Outcome: Serum Testosterone Recovery (>=150 ng/dL) at Months 18 and 24
Description: Percentage of participants with serum testosterone recovery (>=150 ng/dL) at Months 18 and 24 were reported. Testosterone recovery was defined as a serum testosterone level greater than or equal to (>=)150 nanograms per deciliter (ng/dL).
Time Frame: At Months 18 and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Apalutamide Plus ADT (Main Study) + Relugolix Followed by Apalutamide Plus Relugolix (Sub Study)
Number analyzed (Participants) | 108
Percentage of participants
  Month 18 | 42.0 [31.9 to 51.7]
  Month 24 | 77.4 [66.6 to 85.1]

5. Secondary Outcome: Sub-study: Number of Participants With Treatment-emergent Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product and it does not necessarily have a causal relationship with the intervention. TEAEs were defined as any AEs with onset or worsening on or after date of first dose of study intervention through the day of last dose in sub-study.
Time Frame: From 1st dose of study intervention (relugolix on Day -14) up to end of sub-study (Day 28)
Population: Safety analysis set included all participants who received at least 1 dose of apalutamide. Data for this outcome measure was not planned to be collected and analyzed for main study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub Study: Relugolix Followed by Apalutamide Plus Relugolix
Number analyzed (Participants) | 12
Participants | 8

ADVERSE EVENTS:
Time Frame: Main study and sub-study combined: From first dose of study drug (Cycle 1 Day 1 for main study and Cycle 2 Day 1 for sub-study [post transition into main study]) up to end of study (Month 36); sub-study alone: From Day -14 up to end of sub-study treatment (Day 28)
Description: Safety analysis set included all participants who received at least 1 dose of apalutamide. Adverse events data were planned to be collected and analyzed for unique sub-study participants alone and for combined population (along with main study after sub-study participants transitioned into main study).
Groups:
- Main Study Plus Sub-study (Post Transition): In main study, participants received apalutamide 240 milligrams (mg; 4 tablets of 60 mg) orally once daily (QD) along with ADT intramuscular or subcutaneous injection from Cycle 1 Day 1 up to Cycle 12. Each cycle was of 28 days. Sub-study participants upon completion of 28-day sub-study treatment were transitioned into the main study from Cycle 2 Day 1 and continued to receive apalutamide with ADT (oral relugolix) and were included in the main study analysis.
- Sub Study Alone (Before Transition): In sub-study, participants received a loading dose of relugolix 360 mg (3 tablets of 120 mg) on Day -14 and then relugolix 120 mg orally QD up to Day 28 and accompanied by apalutamide 240 mg (4 tablets of 60 mg tablets) orally QD from Day 1 up to Day 28. Upon completion of 28-day sub-study, participants were transitioned into the main study from Cycle 2 Day 1.
Arm/Group | Main Study Plus Sub-study (Post Transition) | Sub Study Alone (Before Transition)
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/12
Serious Adverse Events (participants affected / at risk) | 16/108 | 0/12
Other Adverse Events (participants affected / at risk) | 107/108 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Plus Sub-study (Post Transition) (N=108) | Sub Study Alone (Before Transition) (N=12)
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Covid-19 (Infections and infestations) | 2 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of the Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Plus Sub-study (Post Transition) (N=108) | Sub Study Alone (Before Transition) (N=12)
Vertigo (Ear and labyrinth disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 9 | 0
Fatigue (General disorders) | 58 | 1
Covid-19 (Infections and infestations) | 19 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 0
Dizziness (Nervous system disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 8 | 0
Haematuria (Renal and urinary disorders) | 6 | 0
Pollakiuria (Renal and urinary disorders) | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 23 | 1
Hot Flush (Vascular disorders) | 74 | 4
Hypertension (Vascular disorders) | 8 | 1
Anxiety (Psychiatric disorders) | 6 | 1
Headache (Nervous system disorders) | 6 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application..

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT04523207/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT04523207/SAP_001.pdf